CLINICAL TRIAL: NCT00513136
Title: A Randomized Trial to Evaluate a Family-focused Mind Body Medicine Intervention to Reduce Fatigue Among Breast Cancer Survivors
Brief Title: Fatigue Intervention Trial for Breast Cancer Survivors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mercy Medical Center (Other)
Responsible Party: Principal Investigator, Michael Mullen, Administration, Mercy Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC2007-46
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Fatigue
Keywords: Fatigue; Breast Cancer; Behavioral Research; Quality of Life
MeSH Terms: conditions — Fatigue; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator): 10 week group-based mind body medicine intervention
  Interventions: Behavioral: Group based mind body medicine intervention
- II (Experimental): Group-based mind body medicine intervention with a family focus
  Interventions: Behavioral: Group-based mind body medicine intervention + family focus

INTERVENTIONS:
Behavioral: Group based mind body medicine intervention — Small groups of women (5-15) will participate in 10 weekly sessions that will include learning relaxation and yoga techniques, principles of exercise and nutrition, cognitive behavioral therapy and exploration of common issues and concerns
  Arms: I
Behavioral: Group-based mind body medicine intervention + family focus — In addition to the 10 weekly group-based sessions, women and their key family members will meet twice with a cognitive therapist and family members will participate in selected aspects of the 10 week program.
  Arms: II

SUMMARY:
Thirty to forty percent of breast cancer survivors suffer from persistent fatigue lingering months to years after adjuvant therapy is completed. Although researchers have developed some effective interventions (exercise or group-based holistic program) to treat fatigue, none have addressed the role of the family in the patient's long-term recovery.

The investigators hypothesize that a family-focused intervention in combination with a mind-body group intervention will be more effective in reducing fatigue, improving quality of life, and enhancing family relationships for breast cancer survivors than a group intervention with an individual focus.

DETAILED DESCRIPTION:
We propose to address the persistent fatigue experienced by brest cancer survivors by using a 10 week group-based mind body medicine intervention that includes the family in the process. We believe that this family-centered approach can facilitate better communication, create shared illness experience and relieve conflict. Reducing this pervasive source of stress will not only reduce the survivor's fatigue, but also foster an opposite family dynamic with positive effects in many other aspects of post-treatment recovery. We will compare the effectiveness of a 10 week group intervention to a 10 week group intervention that includes a family focus.

Breast cancer survivors with moderate to severe fatigue will be randomly assigned to one of the two groups and we will measure change in fatigue, quality of life, mood and social support from baseline to end-of-program and then two and six months after program completion.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III Breast Cancer
* At least 3 months since last breast cancer treatment (excluding hormonal therapy or Herceptin).
* 4 week history of persistent moderate to severe fatigue
* Competent to sign informed consent
* Willing to be randomized

Exclusion Criteria:

* Metastatic breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Fatigue | Change from baseline to end-of-intervention and 2 and 6 months post-intervention

SECONDARY OUTCOMES:
Quality of Life; Mood; Social Support | Change from baseline to end-of-intervention and 2 and 6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kathy J Helzlsouer, MD, MHS, Principal Investigator — Mercy Medical Center; Julianne Oktay, PhD, MSW, Principal Investigator — University of Maryland School of Social Work
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States